CLINICAL TRIAL: NCT04222244
Title: Musculoskeletal Neck Impairment in Headaches Attributed to Rhinosinusitis
Brief Title: Musculoskeletal Impairment in Headaches Attributed to Rhinosinusitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Des Moines University (Other)
Collaborators: Texas Tech University (Other); University of Hartford (Other); Youngstown State University (Other); American Academy of Orthopaedic Manual Physical Therapists (Other)
Responsible Party: Sponsor
Other Study IDs: DesMoinesU
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Headache
Keywords: Headache Attributed to Rhinosinusitis; Neck Pain; Musculoskeletal; Cervical; Joint Laxity; Range of Motion; Segmental Mobility; Sinus Headache
MeSH Terms: conditions — Headache; Neck Pain; Joint Instability | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Headache Attributed to Rhinosinusitis Group (HAR): No interventions will be provided.
  Interventions: Other: No intervention will be administered. We are only performing tests and measures.
- Headache-Free Control Group (Control): No interventions will be provided.
  Interventions: Other: No intervention will be administered. We are only performing tests and measures.

INTERVENTIONS:
Other: No intervention will be administered. We are only performing tests and measures. — No intervention will be administered. We are only performing tests and measures.

SUMMARY:
Neck pain, neck muscle weakness, and limited neck range of motion have been shown in individuals with sinus headaches. Individuals in this previous study self-diagnosed their sinus headaches. It is unknown whether or not individuals who have been diagnosed with sinus headaches according to diagnostic criteria also present with musculoskeletal impairments.

The purpose of this study is to determine if musculoskeletal neck impairments are present in individuals diagnosed with headaches attributed to rhinosinusitis compared to people without headaches.

Upper cervical range of motion can be measured using different tests. The side bend rotation test has been suggested as potentially more useful than the flexion rotation test in individuals with hyper-laxity, however, has not been examined in a symptomatic population.

A secondary purpose is to compare the side bend rotation test to the cervical flexion rotation test in people with varying degrees of joint laxity.

DETAILED DESCRIPTION:
Design: Observational, case control Background: A recent study showed neck pain, neck muscle weakness, and limited neck range of motion in individuals who reported having sinus headaches. These impairments are also associated with cervicogenic headaches (headaches originating in the neck), but had not previously been shown in people with sinus headaches.

Because the individuals in this previous study self-diagnosed their sinus headaches, it is possible that they did not have sinus headaches but rather had a different kind of headache. It is unknown whether or not individuals who have been diagnosed with sinus headaches according to diagnostic criteria also present with musculoskeletal impairments.

Purpose 1: The purpose of this study is to determine if musculoskeletal neck impairments are present in individuals diagnosed with headaches attributed to rhinosinusitis (sinus headaches) compared to people without headaches. Question: Do people with diagnosed with headaches attributed to rhinosinusitis have neck pain or impairments in neck strength, neck range of motion, or segmental neck joint mobility compared to people without headaches?

Background for question 2: Upper cervical range of motion can be measured using the flexion-rotation test or the side bend rotation test. The side bend rotation test has been suggested as potentially more useful in individuals with hyper-laxity, however, has not been examined in a symptomatic population.

Purpose 2: To compare the side bend rotation test to the cervical flexion rotation test and manual joint assessment in people with varying degrees of joint laxity. Question: What is the diagnostic accuracy of the side bend rotation test compared to the index tests of the flexion rotation test and manual joint assessment?

ELIGIBILITY:
Inclusion criteria for the headache attributed to rhinosinusitis (HAR) group:

* HAR has been present for at least 12 weeks OR
* Participant has had at least 4 HAR over the past 12 months without persistent symptoms between (chronic or recurrent)
* Diagnosis of headache attributed to rhinosinusitis (or sinus headaches) according to International Classification of Headache Disorders (ICHD-3)

Exclusion criteria for the HAR group:

* History of surgery to the cervical spine
* Whiplash injury within the past 5 years or any persistent symptoms attributable to a whiplash associated disorder
* Diagnosis of any headache type other than sinus headache with exception of an occasional, mild headache for which they have not sought medical care.

Exclusion criteria for the non-headache group (NHA):

* Any history of headaches for which they have sought medical care

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: community sample including community members seen in physical therapy clinics where data collection will occur.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
range of motion | Day 1
  measured with a cervical range of motion device (CROM)

SECONDARY OUTCOMES:
Pain Level | Day 1
  visual analogue scale
disability | Day 1
  Neck Disability Index (self-report questionnaire)
headache impact | Day 1
  Headache Impact Test (self-report questionnaire)
sino-nasal outcome test (SNOT-22) | Day 1
  self-report questionnaire
Cervical side bend rotation test | Day 1
  neck range of motion side bending first, then rotating the head and neck
cervical flexion rotation test | Day 1
  neck range of motion flexing first, then rotating
segmental joint mobility | Day 1
  manual segmental joint examination
neck flexor endurance | Day 1
  neck flexor muscle endurance test in supine
Beighton score | Day 1
  a series of range of motion tests to measure hyper-laxity of joints

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Petersen, PT, Principal Investigator — Des Moines University
Locations (7):
- United States (7):
  - University of Hartford, Hartford, Connecticut
  - Des Moines University, Des Moines, Iowa
  - Performance Rehabilitation, Lafayette, New Jersey
  - Performance Rehabilitation, Totowa, New Jersey
  - Youngstown State University, Youngstown, Ohio
  - The Corvallis Clinic, Corvallis, Oregon
  - Pain Relief and Physical Therapy, Havertown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided